CLINICAL TRIAL: NCT02945696
Title: Abdominal Wall Nerve Blockade: A Comparison With Local Port Site Injection as Well as Between the Use of Ultrasound and Laparoscopy to Guide Placement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: Marcus Malek (Other)
Responsible Party: Sponsor-Investigator, Marcus Malek, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO16050059
Record Dates: First submitted 2016-10-10; First posted 2016-10-26 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Pain
Keywords: nerve block; laparoscopy; anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Local port site injection (No Intervention)
- Ultrasound-guided nerve blocks (No Intervention)
- Laparoscopic guided nerve blocks (Experimental): These patients will receive the same volume of local anesthetic as those in the ultrasound-guided arm, but the delivery of the local anesthetic will be guided by laparoscopy.
  Interventions: Procedure: laparoscopic guided nerve blocks; Drug: Ropivacaine

INTERVENTIONS:
Procedure: laparoscopic guided nerve blocks — It is common to use ultrasound to define the correct plane for abdominal wall nerve blocks, however, the utilization of laparoscopy to identify this plane is a new intervention that is previously undescribed in children.
  Arms: Laparoscopic guided nerve blocks
Drug: Ropivacaine — Ropivacaine is a local anesthetic used to prevent pain during and after procedures. In this study, ropivacaine will be injected either directly at the port sites, or for a regional abdominal wall nerve block, either under ultrasound or laparoscopic guidance.
  Arms: Laparoscopic guided nerve blocks

SUMMARY:
The investigators will perform a prospective randomized study to compare the effectiveness of laparoscopic-guided abdominal wall nerve blocks with local wound site infiltration and with ultrasounded guided abdominal wall blocks.

DETAILED DESCRIPTION:
Pain control after abdominal surgery in children is often a complex, multifaceted problem that requires a multimodal approach to treatment. Infiltration of wounds with long-acting local anesthetic, either into the surgical field or through locoregional nerve blockade, has been known to decrease narcotic requirements. Nerve blocks of the abdominal wall can occur through several modalities, among them the transverse abdominis plane block and the rectus sheath block. The transversus abdominis plane (TAP) block places local anesthetic in a plane between the internal oblique and transversus abdominis muscles, directly blocking innervation of spinal nerves T9-L3, the ilioinguinal, iliohypogastric and lateral cutaneous branches of L1-3, reducing pain sensation to the anterior abdominal wall. The rectus sheath block places local anesthetic between the internal oblique and transversus abdominis at the level of the terminal branches of intercostal nerves 9-11.

The investigators will perform a prospective randomized study to compare the effectiveness of laparoscopic-guided abdominal wall nerve blocks with local wound site infiltration and with ultrasounded guided abdominal wall blocks.

The goal of this study is to determine whether patients who receive a nerve block have significantly less pain compared to patients who receive local infiltration of anesthetic. Secondly, the investigators believe that laparoscopic-guided abdominal wall nerve blocks should be as effective as abdominal wall blocks performed under ultrasound-guidance, and may in fact allow for more consistent infiltration of local anesthetic to desired nerve bundles. Thirdly, the investigators believe that laparoscopic-guided abdominal wall nerve blocks are significantly less time intensive than ultrasound-guided abdominal wall nerve blocks, allowing a cost savings and decreased time under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 5 - 17 years old.
2. Patients undergoing laparoscopic procedures
3. Patients that weigh greater than or equal to 34 kg and less than 100 kg.

Exclusion Criteria:

1. Patients who underwent open surgical procedures will be excluded from this study.
2. Patients that weigh less than 34kg.
3. Patients that weigh more than 100 kg.
4. Perforated appendicitis.
5. Bowel obstruction

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Minutes under anesthesia | 2 years

SECONDARY OUTCOMES:
Pain scores | 2 years
Narcotic usage | 2 years

IPD SHARING:
Plan to Share IPD: No